CLINICAL TRIAL: NCT03362671
Title: Bimaxillary Implant Supported Mandibular Advancement Pilot
Brief Title: Implant Supported Oral Appliance Treatment of OSA
Acronym: BIMA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the initial design of the novel oral appliance proved uncomfortable and thus terminated trial after three subjects.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Benjamin Pliska, Assistant Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14G31862
Record Dates: First submitted 2017-11-23; First posted 2017-12-05 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Mandibular Advancement Splint; Oral Appliance; Treatment; Orthodontic Implants
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Participants will be treated with a novel experimental implant supported mandibular advancement oral appliance, which uniquely attaches to orthodontic mini implants (OMIs) in the jaw. Participants will be fitted with OMIs per standard clinical practice prior to treatment with the novel oral appliance.
  Interventions: Device: Implant Supported Mandibular Advancement Oral Appliance; Device: Orthodontic Mini Implant

INTERVENTIONS:
Device: Implant Supported Mandibular Advancement Oral Appliance — This device is a novel oral appliance that attached to orthodontic mini implants in the jaw and is designed to keep the jaw in an advanced position, opening the upper airway during sleep.
Device: Orthodontic Mini Implant — Small titanium devices that are fixed to the bone for the purpose of enhancing anchorage of other orthodontic devices.
  Other Names: Temporary Anchorage Devices (TADs)

SUMMARY:
Mandibular advancing oral appliances (OAm) are an effective and increasingly common treatment modality for the management of obstructive sleep apnea (OSA) in adults.

The effectiveness of OAm therapy, however, is dependent on a high level of patient adherence, which may be negatively impacted by treatment side effects - the most significant of which are occlusal changes and tooth movement.

The proposed pilot study will evaluate the efficacy of a novel implant supported OAm in 10 OSA patients who have already been successfully treated with a traditional OAm.

The study will compare OSA specific outcomes with traditional OAm use against novel oral appliance use after one month. This study could potentially validate the novel design features of an effective treatment option for OSA that does not result in tooth movement, which is a significant side effect shared by all existing OAm devices.

Ultimately, this study could lead to increased treatment adherence and better OSA patient health outcomes in the future.

DETAILED DESCRIPTION:
Mandibular advancement oral appliances (OAm) are devices that keep the airway open during sleep by pulling the lower jaw forward. OAm have been shown to be an effective treatment for both mild and severe OSA. OSA is a chronic disease and there is no cure. OSA treatments depend on high patient adherence for long term effectiveness.

Currently marketed OAm devices attach to the teeth as a way of holding the jaw in position. However, attaching directly to the teeth causes unwanted tooth movement with long term OAm use. As a result, some long-term users of OAm have stopped treatment due to a decrease in quality of life caused by tooth movement. Accordingly, the changes in tooth position can be seen as a limitation of the existing appliances. For this reason, there is a strong need for a type of treatment that can effectively pull the jaw forward without causing movement of the teeth, which is inevitable with the way the current OAm devices work.

This trial is a pilot study to find out if a novel OAm device is an effective treatment for OSA. The novel OAm device does not contact the teeth directly but instead attaches to orthodontic mini implants (OMIs) in the jaw. 10 OSA patients who have previously been successfully treated with a traditional OAm appliance will be fitted with the novel oral appliance. Participants will be fitted with 6 OMIs following standard practice and the bespoke oral appliance will be manufactured and delivered to the patient for use.

Prior to receiving treatment, participants will undergo a baseline assessment where demographic, anthropometric, and specific periodontal health data will be collected. Daytime sleepiness will be assessed and at-home sleep test will be used to establish baseline sleep parameters with the existing appliance.

Follow up sleep tests will be completed 1 month after initiation of treatment with the new appliance. ESS questionnaires and treatment experience interviews will be completed at 1 month and 4 months after the start of treatment with the new appliance. Treatment adherence and OMI side effects will be monitored throughout the study. Patients will be given the option of continuing treatment with the novel device or having the implants removed and returning to treatment with their previous OAm.

To directly address the primary aim of this study, OSA related parameters will be measured by a combination of methods including at-home sleep tests and Epworth Sleepiness Scale (ESS) questionnaires. Secondary outcome variables to assess treatment adherence and satisfaction include self-reported adherence data using sleep diaries, experience interviews and assessing OMI side effects throughout the study.

ELIGIBILITY:
Inclusion Criteria:

This trial will recruit 10 patients with an objective diagnosis of obstructive sleep apnea who are not naïve to treatment. The inclusion criteria are:

* Currently receive or have previously received successful OSA treatment with an OAm;
* Age 25 - 65 years old, who are able to freely provide informed consent;
* Body Mass Index (BMI) ≤ 35;
* Apnea-Hypopnea Index (AHI) within the range 5≤AHI≤50 documented with polysomnography in the last 2 years ***OR***
* Respiratory Disturbance Index (RDI) within the range 20 ≤ RDI ≤ 50 documented with Level III portable sleep test ***OR***
* Oxygen Desaturation Index (ODI) ≥ 10

Exclusion Criteria:

The patient is excluded if it meets any of the following criteria:

* Extensive periodontal disease;
* Bleeding disorder;
* Bone metabolic disorder
* Immunocompromised
* Diabetes mellitus
* Xerostomia
* Titanium allergy
* Insufficient vertical opening to accommodate treatment with OAm;
* Pregnancy (if a participant becomes pregnant during the trial, the participant will be withdrawn from the study).
* Uncontrolled congestive heart failure (defined as a prior clinical diagnosis, an ejection cut-off of 40% or clinical sign in the opinion of a primary care physician or cardiologist) that makes it unsafe in the opinion of the investigators for the subject to participate in the trial;
* Coronary artery disease unless stable for at least 6 months and considered by the investigators to have a stable disease;
* Any history of angina, myocardial infarction or stroke;
* Any history of major depressive disorder along with current moderate-severe disease;
* Active cancer management (unless in remission for more than 1 year);
* Known renal failure (with need for dialysis)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea Index (AHI) | Data collected at 0, and 1 months after initiation of treatment with the new appliance.
  Indication of the severity of sleep apnea. The AHI is calculated by dividing the number of apnea events by the number of hours of sleep. This outcome will assess the change in AHI over time.

SECONDARY OUTCOMES:
Daytime Sleepiness | Data collected at 0, 1, and 4 months after initiation of treatment with the new appliance.
  Evaluation of OSA specific fatigue using Epworth Sleepiness Scale (ESS) questionnaire. ESS measures daytime sleepiness via 8 questions that ask about daytime sleepiness during common everyday conditions. The potential range of scores for any questions is from 0 to 3. Higher values represent worse outcomes. Their are no subscales for ESS. The answers to the questions are all summed up. Total score ranges between 0 and 24. A score above 10 indicates daytime sleepiness with higher scores indicating more sleepiness.
Arterial Oxygen Saturation | Data collected at 0, 1, and 4 months after initiation of treatment with the new appliance.
  Using a pulse oximeter to determine the percentage of hemoglobin binding sites in the bloodstream occupied by oxygen.
Treatment Adherence | Data will be collected by the research team 4 months after initiation of treatment with the new appliance.
  Self-reported use of the appliance by recording the number of hours per night and the number of nights per week that the appliance is used.
Patient Experience | Data collected 1 and 4 months after initiation of treatment with the new appliance.
  Subjective patient experience data collected from semi-structured interviews.
Mini Implant Side Effects - Mobility | Data collected at 1 week, 1 month and 4 months after initiation of treatment with the new appliance.
  Using tactile assessment to determine implant mobility per Ngiam et al. Mobility will be graded from 0-2 depending on severity. 0 represents no mobility whereas 2 represents mobility greater than 1mm. There is an additional option for total mobility or implant loss.
Mini Implant Side Effects - Gingival Irritation | Data collected at 1 week, 1 month and 4 months after initiation of treatment with the new appliance.
  Gingival irritation will be determined using tactile/visual assessment. Irritation will be scored as either YES (present) or NO (absent).
Mini Implant Side Effects - Soreness | Data collected at 1 week, 1 month and 4 months after initiation of treatment with the new appliance.
  Soreness will be determined using tactile/visual assessment and self-reported by patients. Soreness will be scored as either YES (present) or NO (absent).
Mini Implant Side Effects - Jaw Pain | Data collected at 1 week, 1 month and 4 months after initiation of treatment with the new appliance.
  Jaw pain will be determined using tactile/visual assessment and self-reported by patients. Jaw pain will be scored as either YES (present) or NO (absent).
Mini Implant Side Effects - Excess Salivation | Data collected at 1 week, 1 month and 4 months after initiation of treatment with the new appliance.
  Excess salivation will be determined using visual assessment and self-reported by patients. Excess salivation will be scored as either YES (present) or NO (absent).
Mini Implant Side Effects - Other | Data collected at 1 week, 1 month and 4 months after initiation of treatment with the new appliance.
  A brief description of any other side effects will be self-reported by patients.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin T Pliska, DDS, Principal Investigator — University British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada